CLINICAL TRIAL: NCT03738085
Title: Previous Abdominal Surgery and Obesity Does Not Affect Unfavorably the Outcome of Total Laparoscopic Hysterectomy
Status: Completed | Type: Observational
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, Batuhan Turgay, Principal Investigator, Ankara University
Other Study IDs: AnkaraU-12-562-16
Record Dates: First submitted 2018-11-08; First posted 2018-11-13 (Actual); Last update posted 2018-11-14 (Actual); Status verified 2018-11

CONDITIONS: Laparoscopic Surgical Procedure; Obesity; Surgery--Complications
Keywords: Complication; Previous surgery; Total laparoscopic hysterectomy; Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Previous abdominal surgery group: Previous abdominal surgery group underwent total laparoscopic hysterectomy
- No previous abdominal surgery group: No Previous abdominal surgery group underwent total laparoscopic hysterectomy
- Obese patients underwent TAH: BMI≥30 kg/m2
- Obese patients underwent TLH: BMI≥30 kg/m2

SUMMARY:
Previous surgery and obesity has disputed as an unfavorable factor during Total Laparoscopic Hysterectomy. The aim of the investigator's study was to assess the effects of previous abdominal surgery and obesity on intra-operative and post-operative outcomes of TLH.

DETAILED DESCRIPTION:
Abstract:

Objective: To assess the effects of previous abdominal surgery and obesity on the intra-operative and post-operative outcomes of total laparoscopic hysterectomy (TLH).

Method: In this retrospective cohort study, women who underwent TLH for benign conditions between January 2011 and December 2016 in tertiary academic center were included. Patients were grouped according to previous abdominal surgery. The study group consisted of patients who had at least one previous abdominal surgery and the control group consisted of patients with no previous abdominal surgery. In a further analysis, a subgroup of obese patients with BMI (body mass index) ≥30 kg/m2 was evaluated. For this analysis, the obese patients who underwent TLH were picked up and the results were compared to the results of obese patients who underwent total abdominal hysterectomy (TAH) during the same time period. The main outcome parameters were duration of hospital stay and major complication rate.

ELIGIBILITY:
Inclusion Criteria:

* all women who underwent TLH for benign conditions during study period
* all obese ≥30 kg/m2 women who underwent TAH for benign conditions during study period

Exclusion Criteria:

* No

Ages: 35 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — participant eligibility is based on self-representation of gender identity and physical status
Study Population: All women who underwent TLH for benign conditions
Sampling Method: Probability Sample
Enrollment: 380 (Actual)
Dates: Start 2011-01 (Actual); Primary Completion 2014-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Complication rate | Up to one week
  Evaluate the complication number between groups
Hospital stay difference | Up to one week
  Evaluate the difference of hospitalization day between groups

CONTACTS AND LOCATIONS:
Overall Officials: Batuhan Turgay, Principal Investigator — Ankara University; Bulent Berker, Professor, Principal Investigator — Ankara University

IPD SHARING:
Plan to Share IPD: Undecided